CLINICAL TRIAL: NCT06741280
Title: Post-marketing Study for the Evaluation of the Efficacy and Safety of Profilm Mouth Sores
Brief Title: Post-marketing Study for the Evaluation of Profilm Mouth Sores
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: i+Med S.Coop. (Industry)
Collaborators: Dr. Goya Análisis, SL. (Industry); Centro Médico Complutense Grupo Virtus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROFILM AFTAS-PIC01-2022
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Mouth Sores
Keywords: Ulcers; Recurrent aphthous stomatitis; Oral ulcers; Mouth ulcers; Mouth sores; Sore
MeSH Terms: conditions — Oral Ulcer; Ulcer; Stomatitis, Aphthous

STUDY DESIGN:
Intervention Model Description: Post-marketing, prospective, within-subject controlled clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Profilm Mouth Sores (Experimental): To evaluate the efficacy and safety of the Profilm Mouth Sores for the treatment of mouth sores.
  Interventions: Device: Profilm Mouth Sores

INTERVENTIONS:
Device: Profilm Mouth Sores — Daily applications of the product as soon as a mouth sore appears, until its complete disappearance or healing, as follows: application every 8 hours, with the possibility of shortening the interval to 6 hours if needed (a maximum of 3-4 applications).

SUMMARY:
The study aims to assess the effect of Profilm Mouth Sores treatment for relieving symptoms caused by mouth sores. It will involve 35 participants and last around 14 days or until the sores heal, with three daily applications. A dermatology specialist will evaluate the results through tests and examinations of the treated area.

ELIGIBILITY:
Inclusion Criteria:

* Male / female / aged 18 years or older.
* Presence of an ulcer on the oral mucosa, regardless of the number of days since its appearance.
* At least 30 days have passed since the last episode.
* Willingness to return for all study-related visits.
* Sufficient willingness and ability, as judged by the investigator, to respond to the questionnaires included in the study.

Exclusion Criteria:

* Pregnant women or women in the breastfeeding period.
* Patients undergoing treatment with antiviral medications, hydrocortisone, or other medications.
* Patients with immunodeficiency diseases, such as acquired immunodeficiency syndrome or altered immune activity in the last 7 days.
* Patients undergoing other pharmacological therapy for oral conditions.
* Patients with other oral mucosa diseases simultaneously.
* Known allergy or hypersensitivity to any of the components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-12-13 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Confirm the effectiveness of the treatment in terms of pain relief, using an EVA scale. | At baseline, in 24 hours, in 3 days, in 7 days and in 14 days.
  For the evaluation of effectiveness, a 0 to 10 EVA scale is used (where 0 = no pain / 10 = severe or unbearable pain).
Serious adverse events. | Through study completion, apprroximately 2 weeks.
  Evaluate the safety of the treatment, in terms of the incidence of serious adverse events.

OTHER OUTCOMES:
Mild adverse events. | Through study completion, apprroximately 2 weeks.
  Evaluate the incidence of other mild and transient adverse events related to the product.
Healin time and lesion size. | At baseline, in 24 hours, in 3 days, in 7 days and in 14 days.
  Reduction in healing time and extent of the ulcer. Mean healing time of the lesion ≤ 14 days or % of patients with complete healing ≥ 70% at one week.
Global treatment assessment by participants. | At the conclusion of the study, approximately 2 weeks later.
  Global treatment assessment questionnaires will evaluate the effectiveness of the treatment on a scale from 0 to 10 (where 0 = no response or not satisfied at all, and 10 = excellent response or exceptionally satisfied).
Number, size, and location of sores | At baseline, in 24 hours, in 3 days, in 7 days and in 14 days.
  Determination of the number, size, and location of sores, as well as difficulty eating and/or drinking.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Médico Complutense Grupo Virtus, Alcalá de Henares, Madrid, Spain